CLINICAL TRIAL: NCT01837563
Title: Monitoring of Neoadjuvant Therapy in Locally-Advanced Breast Cancer
Status: Terminated | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D0605
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Locally Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether four new alternative imaging methods can be used to follow the response of breast cancer to the treatment patients are being given. These methods produce an image of the inside of the breast so that doctors can better decide whether breast cancer is responding to therapy. An important part of the study is to examine the same person with all methods in order to directly compare results. The four methods are: MRI Elasticity Imaging (abbreviated MRE), Electrical Impedance Spectroscopy (abbreviated EIS), Microwave Imaging and Spectroscopy (abbreviated MIS), Near Infrared Spectroscopy (abbreviated NIR). In addition to the experimental imaging methods, patients may also undergo a contrast-enhanced MRI, and/or additional mammography, which will help researchers compare the experimental methods. These additional examinations are accepted diagnostic procedures; they are not experimental. Some participants will have one or both of these additional examinations if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced breast cancer, with or without metastatic disease
2. Patient to receive systemic therapy
3. Breast size and epithelial integrity adequate to allow alternate imaging exams.
4. Patient able to provide written informed consent.
5. No serious associated psychiatric illness
6. Age ≥ 18 years old

Exclusion Criteria:

1. Cardiac pacemaker
2. Any implanted electronic device
3. Severe claustrophobia
4. Allergy to the MRI contrast agent gadolinium

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with locally-advanced breast cancer, with or without metastatic disease, meeting inclusion criteria (and giving informed consent for participation) receiving systemic therapy at DHMC will be enrolled. Breast size and epithelial integrity of the skin surface can limit the ability to deliver effective imaging exams, adn these individual characteristics need be determined in each individual patient. Women with pacemakers or other implanted electronic devices will not be allowed into the study because of potential for electrical interference with proper operation during an imaging session.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Objective Response | at baseline, at conclusion of treatment (up to 6 months)
  Correlate changes in each imaging modality with objective response to therapy, as defined by conventional criteria (clinical exam and conventional imaging).

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States